CLINICAL TRIAL: NCT03064711
Title: Comparison of Activity and Fatigue of the Respiratory Muscles and Pulmonary Characteristics Between Post-Polio Patients and Healthy Controls: A Pilot Study
Brief Title: Activity and Fatigue of the Respiratory Muscles and Pulmonary Characteristics in Post-Polio Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Isabella Shvartz, MD, Hadassah Medical Organization
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Tali- HMO-CTIL
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Post-polio Syndrome
MeSH Terms: conditions — Postpoliomyelitis Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electronyugraphy — Surface electromyography (sEMG) recorded diaphragmatic muscle activity during rest and while performing maximal voluntary ventilation

SUMMARY:
Background: Early diagnosis of respiratory impairment in Post-Polio (PPS) patients may delay respiratory decline and future need of invasive respiratory aids.

Objectives: To compare pulmonary function measures, maximal respiratory pressure and activity levels and fatigue of respiratory muscles between patients with PPS and healthy controls.

Design: Cross-sectional study. Setting: Hadassah physical medicine and rehabilitation department, Jerusalem. Patients: Patients with PPS (N=12; 6 males; age 62.1±11.6 years) able to walk for 6 minutes without human assistance; age-matched healthy subjects (N=12; 4 males; age 62.2±6.5 years).

Intervention: None. Measurements: A body plethysmograph was used to quantify forced expiratory volume in the first second of a forced expiratory maneuver, vital capacity, slow vital capacity, Residual Volume (RV), Total Lung Capacity (TLC), and Thoracic Gas Volume (TGV). Also, RV to TLC ratio is calculated. A manometer was used to measure Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP). A spirometer was used to measure Maximal Voluntary Ventilation (MVV). Surface electromyography (sEMG) recorded diaphragmatic muscle activity during rest and while performing MVV.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with post-polio syndrome
* Able to walk for 6 minutes, with or without walking aids and orthotics but without human assistance

Exclusion Criteria:

* Any neurological or orthopedic condition, unrelated to post-polio syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Median frequency of electromyography | Two hours
  measure related to fatigue measured during maximal voluntary ventilation

SECONDARY OUTCOMES:
Pulmonary function | Two hours
  Measured using a body plethysmograph
maximal inspiratory/expiratory pressures | Two hours
  Measured using ahand-held portable, digital manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel